CLINICAL TRIAL: NCT02320019
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 2b Trial to Evaluate the Efficacy and Safety of YH14618 in Patients With Lumbar Degenerative Disc Disease
Brief Title: Clinical Trial of YH14618 in Patients With Degenerative Disc Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YH14618-202
Record Dates: First submitted 2014-12-11; First posted 2014-12-19 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Disc Degenerative Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Group A (Experimental): YH14618 A mg/disc
  Interventions: Drug: YH14618
- Group B (Experimental): YH14618 B mg/disc
  Interventions: Drug: YH14618
- Group C (Experimental): YH14618 C mg/disc
  Interventions: Drug: YH14618
- Group D (Experimental): YH14618 D mg/disc
  Interventions: Drug: YH14618

INTERVENTIONS:
Drug: Placebo — Placebo matching YH14618
  Arms: Placebo group
Drug: YH14618
  Arms: Group A; Group B; Group C; Group D

SUMMARY:
Research Hypothesis:

There will be a greater proportion of VAS responders defined as those who achieve ≥ 50% reduction from baseline in VAS for low back pain at week 12 following intradiscal injection of YH14618 compared to placebo. Patients have been diagnosed as one or two symptomatic lumbar degenerative disc disease defined as Pfirrmann grade 2 to 4 using MRI. Patients have suffered from persistent low back pain with at least 3 months of conservative therapy and must have low back pain measured by VAS≥4 cm and modified Oswestry disability index (mODI) ≥30% at the baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as one or two symptomatic early lumbar (L1/L2 ~ L5/S1) degenerative disc disease defined as Pfirrmann grade 2 to 4 using MRI performed within 4 weeks prior to randomization.
* Patients have suffered from persistent low back pain with at least 3-month conservative therapy.
* Patients have low back pain measured by VAS≥4cm and mODI≥30% at screening and randomization visit (Day 0).

Exclusion Criteria:

* Clinically significant spine compression fracture, spinal stenosis, or spinal instability.
* Clinically significant sacroiliac joint dysfunction, facet joint pain, or those who are suspected.
* Modic change type III assessed by X-ray and MRI
* History of spine surgery
* Neurologic disorders.
* Any other systemic disease which can influence spine such as rheumatoid arthritis, ankylosing spondylitis, or autoimmune disease.
* Participation in other clinical trials with intradiscal injection (eg, Phase 1/2a YH14618-201 trial, or Cell therapy, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Proportion of VAS responders | at 12-week
  Proportion of VAS responders defined as those who achieve ≥ 50% reduction in VAS at week 12 from baseline

SECONDARY OUTCOMES:
Proportion of VAS responders | at 24-week
Proportion of mODI responder | at 12-week, 24-week
Changes in VAS score from baseline | Each visit for 24 weeks
Changes in mODI score from baseline | Each visit for 24 weeks

OTHER OUTCOMES:
Proportion of moderate VAS responder | at 12-week, 24-week
  Moderate VAS responder are defined as those who achieve ≥ 30% reduction in VAS from baseline
Percent change from baseline to Week 12 and 24 for VAS | Each visit between Week 12 and 24
Proportion of patients who are being VAS responders at Week 12 and maintain the treatment effect of ≥ 50% reduction in VAS up to week 16, 20, and 24 | Each visit between Week 12 and 24
Proportion of patients who are being mODI responders at Week 12 and maintain the treatment effect of ≥ 15 points reduction in mODI up to week 16, 20, and 24 | Each visit between Week 12 and 24
Change in VAS from Week 12 to Week16, 20, and 24 | Each visit between Week 12 and 24
Change in mODI from Week 12 to Week 16, 20, and 24 | Each visit between Week 12 and 24
Time to achieve the first ≥ 50% reduction in VAS following the intradiscal injection of Investigational product | For 24 weeks
Pfirrmann grade using MRI at Week 24 | Screening, Week 24
Percent change from baseline to Week 24 for Disc Height Index (DHI) | Screening, Week 24
Quality of life measured by EQ-5D and SF-12 | at Week 12 and 24
Quality of life measured by EQ-5D | at Week 12 and 24
Quality of life measured by SF-12 | at Week 12 and 24
Patient global impression of change | at Week 12 and 24
Clinical global impression of change | at Week 12 and 24
Time to analgesic rescue following the intradiscal injection of Investigational product | For 24 weeks
Amount of rescue medication tablets taken following the intradiscal injection of Investigational product | For 24 weeks
The number of days taken rescue medication following the intradiscal injection of investigational product | For 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Su Youn Nam, M.D., Ph.D., Study Director — Yuhan Corporation
Locations (1):
- Severance Hospital, Seoul, South Korea